CLINICAL TRIAL: NCT04819477
Title: Can Austrian Lung Specialists' Assessments of Lung Cancer Screening be Influenced by a Fact Box?"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Landsteiner Institute for Lung Research and Pneumological Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Version 5.0. / 14.10.2020
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cate Plots (Other): after being asked about current referral practices and assessment of benefits and risks of lung cancer screening, all respondents will receive the Fact box after which they will be randomized into two equal groups. The first group (Arm 1) receives a Cates plot and then another survey about assessment of benefits and risks of lung cancer screening and potential change in referral behavior.
  Interventions: Behavioral: Fact box; Behavioral: Cates plot
- Fact box only (Other): after being asked about current referral practices and assessment of benefits and risks of lung cancer screening, all respondents will receive the Fact box after which they will be randomized into two equal groups. The second group (Arm 2) receives then a survey about assessment of benefits and risks of lung cancer screening and potential change in referral behavior
  Interventions: Behavioral: Fact box

INTERVENTIONS:
Behavioral: Fact box — All physicians surveyed receive a fact box with numerical information on the benefits and harms of chest CT as a screening method.
  In addition to the fact box, half of the participants will be randomly assigned to receive the same information in the form of a Cates plot.
Behavioral: Cates plot — In addition to the fact box, half of the participants will be randomly assigned to receive the same information in the form of a Cates plot.
  Arms: Cate Plots

SUMMARY:
Lung cancer is the most frequently dianosed cancer worldwide. To date, no screening method has been able to establish itself as routinely recommended by the guidelines. In this prospective study with 1:1 randomized questioning using an Internet tool, physicians will be asked in 2 phases (before and after intervention with a fact box) about their assessment of the benefits and risks of lung cancer screening by thoracic computed tomography and about a potential intention to change referral behavior. Randomly assigned, half of the participants will receive the same information in addition to the fact box graphically presented as a Cates plot.

DETAILED DESCRIPTION:
The topic of lung cancer screening is highly topical and relevant in that this cancer is the most frequently diagnosed worldwide and has the highest mortality among malignancies. To date, no screening method has been able to establish itself as routinely recommended by the guidelines. In the recently published Dutch-Belgian NELSON study on low dose thoracic CT as a screening method in high-risk patients (smokers and ex-smokers), an - albeit small - reduction in mortality was shown in the screening group vs. the control group).

A prerequisite for a detailed information of the patient about the implementation as well as the advantages and disadvantages of screening is that the physician has risk competence and knows and is able to interpret the screening data. The use of a fact box can be used to improve knowledge of statistical data.

In this prospective study with 1:1 randomized questioning using an Internet tool, physicians will be asked in 2 phases (before and after intervention with a fact box) about their assessment of the benefits and risks of lung cancer screening by thoracic computed tomography and about a potential intention to change referral behavior. Randomly assigned, half of the participants will receive the same information in addition to the fact box graphically presented as a Cates plot.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Austrian Society of Pneumology (ÖGP) with a completed pulmonary subject and members of the Austrian Radiological Society (ÖRG), Society for Medical Radiology and Nuclear Medicine with a completed subject.

Exclusion Criteria:

* Non members of the Austrian Society of Pneumology (ÖGP)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
CT-Screening | through study completion, an average of 1 year
  Proportion of physicians CT-Screening

CONTACTS AND LOCATIONS:
Overall Officials: Georg-Christian Funk, MD, Principal Investigator — 2nd Medical Department with Pneumology
Locations (1):
- Karl Landsteiner Institut für Lungenforschung und Pneumologische Onkologie, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No